CLINICAL TRIAL: NCT01960270
Title: Secondary Bilateral or Controlateral Sacral Nerve Stimulation in Overactive Bladder Patients With Unilateral Stimulation Failure - Multicenter Study
Brief Title: Secondary Bilateral Sacral Nerve Stimulation in Overactive Bladder Patients
Acronym: NEUROBIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/003/HP
Record Dates: First submitted 2013-07-04; First posted 2013-10-10 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Bladder Hyperactivity
Keywords: relapse after an initial clinical response
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alone controlateral stimulation (Experimental): Device: INTERSTIM II
  * Stimulator II activated
  * Stimulator I not activated
  * Measure of efficacy on bladder hyperactivity
  Interventions: Device: Device: INTERSTIM II
- 2 sides-stimulation (Experimental): Device: INTERSTIM II
  * Stimulator I and II activated
  * Measure of efficacy on bladder hyperactivity
  Interventions: Device: Device: INTERSTIM II

INTERVENTIONS:
Device: Device: INTERSTIM II — A second stimulator is implanted on controlateral site

SUMMARY:
Unilateral sacral neuromodulation (SNM) has emerged as a valuable treatment for patient with low urinary tract dysfunction when failure or bad tolerance to anticholinergic treatment for overactive bladder. However, in the medium or long term, some patients failed to benefit from unilateral stimulation (unilateral neuromodulation). A contralateral stimulation could be tested then implanted to restore the efficacy. An other option is to perform a bilateral stimulation of the sacral nerves that could lead to a summation effects better than unilateral stimulation. Therefore, if a unilateral sacral nerve stimulation fails, a contralateral or a bilateral test should be considered.

DETAILED DESCRIPTION:
Sacral neuromodulation (SNM) is a treatment in non neurogenic (idiopathic) patients with overactivity of the bladder (OAB) symptoms, refractory to conservative treatment. After selection of patients with positive stimulation test (PNE test), the success rate of stimulation implant is approximatively 70% (40 to 80%). Unilateral versus bilateral initial implantation was retrospectively compared by Pham et al. with respectively 58 and 77% success rate. Wound infection and complication rate were similar. However the limitation of bilateral stimulation is an increased cost for the health care system, augmented duration of the procedure, possible morbidity. Therefore initial implantation in the first step of the treatment is unilateral in current practice. However, after a period of time, a secondary failure may happen, either a complete failure with return to initial symptom or a partial failure with a decrease of the efficacy that may impact on quality of life. However, a non clinical evident effect could have a summation effect if a contralateral stimulator was implanted, and possibly better than contralateral alone.

Research have shown in a small study on 15 patients that a selected group of patients appear to benefit from bilateral stimulation test (PNE test) after failure of unilateral S3 stimulation. A successful response was observed in 4/11 (36%) OAB patients. Bilateral stimulation induced a higher clinical response than stimulation of a controlateral lead alone in voiding parameters. In the patients who showed a successful response to PNE test, 3 were implanted bilaterally with more than 50% improvement for 2 of them at one year follow-up, and 41% improvement for the third. No painful stimulation or side effects were reported with chronic bilateral stimulation. In one study, a lead migration was suspected in 3/15 patients and was the cause of failure. Therefore the proposed study will use systematically a tined lead electrode that avoid lead migration.

According to these preliminary data, test stimulation with a contralateral lead might be considered in secondary unsuccessful patient and evaluated. Further investigation is necessary to determine in a larger cohort the result of contralateral alone or bilateral stimulator implantation. There is no established guidelines in secondary unsuccessful patients, therefore contralateral stimulation is used in clinical practice according to patient and practitioner opinion. This protocol is presented as a standard clinical practice evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with Sacral Neuro Modulation for idiopathic OAB with initial efficacy of at least 3 months following by a failure despite optimization of the stimulation (minimum 3)
* OAB evaluated by voiding diary: number of frequency ≥ 8/24 h or urgencies ≥ 3 during 3 days, with or without urge incontinence.
* Age between 18 and 80 years.

Exclusion Criteria:

* Psychiatric or neurologic disabilities on neurologic evaluation.
* Bladder lithiasis or tumor (cystoscopy or ultrasonography).
* Treatment by drugs that could interfere with the OAB syndromes.
* Pelvic floor exercises should have been interrupted 1 month before.
* No planned surgery on bladder or urinary neurologic tract.
* Diuresis > 3 liters per 24 hours.
* Negative test at the end of screening period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Success of Test Period | Day 0
  A successful response is defined as greater than 50% improvement in at least one relevant voiding parameters, with bilateral stimulation versus baseline without stimulation. Relevant voiding diary parameters are: urgency number, frequency, urge incontinence number. These criteria are commonly used in the studies on sacral neuromodulation.

SECONDARY OUTCOMES:
Effect of alone controlateral stimulation | Day 30 and day 60
  Effect of alone controlateral stimulation on : urgency, frequency, urge incontinence.
Effect of alone controlateral stimulation | Day 30 and day 60
  Effect of alone controlateral stimulation on : Quality of Life (QoL) scores
Effect of alone controlateral stimulation | Day 30 and day 60
  Effect of alone controlateral stimulation on : VAS pain scale
Effect of alone controlateral stimulation | Day 30 and day 60
  Effect of alone controlateral stimulation on : Adverse events.
Effect of alone controlateral stimulation | Day 30 and day 60
  Prognostic factors of success will be evaluated concerning age, sex, urodynamic parameters, period of time of symptoms before first implant, period of time between first implant and controlateral/bilateral stimulation, complete failure or a partial failure of efficiency of initial stimulator.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GRISE, Pr, Principal Investigator — UH Rouen
Locations (12):
- France (12):
  - UH Caen, Caen
  - UH Grenoble, Grenoble
  - GHICL Lille Saint Philibert, Lille
  - Lille University Hospital, Lille
  - Hospices civiles de Lyon, Lyon
  - AP-HM, Marseille
  - UH Nantes, Nantes
  - UH Nîmes, Nîmes
  - AP-HP Pitié Salpetrière, Paris
  - AP-HP Tenon, Paris
  - UH Rouen, Rouen
  - UH Toulouse, Toulouse

REFERENCES:
- [Result] van Kerrebroeck PE, van Voskuilen AC, Heesakkers JP, Lycklama a Nijholt AA, Siegel S, Jonas U, Fowler CJ, Fall M, Gajewski JB, Hassouna MM, Cappellano F, Elhilali MM, Milam DF, Das AK, Dijkema HE, van den Hombergh U. Results of sacral neuromodulation therapy for urinary voiding dysfunction: outcomes of a prospective, worldwide clinical study. J Urol. 2007 Nov;178(5):2029-34. doi: 10.1016/j.juro.2007.07.032. Epub 2007 Sep 17. PMID 17869298
- [Result] Pham K, Guralnick ML, O'Connor RC. Unilateral versus bilateral stage I neuromodulator lead placement for the treatment of refractory voiding dysfunction. Neurourol Urodyn. 2008;27(8):779-81. doi: 10.1002/nau.20577. PMID 18551562
- [Result] Marcelissen TA, Leong RK, Serroyen J, van Kerrebroeck PE, De Wachter SG. The use of bilateral sacral nerve stimulation in patients with loss of unilateral treatment efficacy. J Urol. 2011 Mar;185(3):976-80. doi: 10.1016/j.juro.2010.10.065. Epub 2011 Jan 19. PMID 21247601